CLINICAL TRIAL: NCT05073445
Title: Stress and Resilience in Anesthesia Professionals
Acronym: ResiStress
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 02021 - 097
Record Dates: First submitted 2021-07-29; First posted 2021-10-11 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Stress, Professional; Resilience; Anaesthesiology; High Fidelity Simulation
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SDNN measurement — SDNN measurement during pediatric simulation

SUMMARY:
The purpose of this study was to analyze the correlation between the resilience of anesthesia professionals and the stress measured during a simulation session.

DETAILED DESCRIPTION:
This trial will be carried out at the simulation center of the training institute for health professionals of the CHU Grenoble Alpes. Volunteer anesthesia professionals and students will perform a scenario simulating a pediatric laryngospasm during a surgical incision.

Each scenario will be performed by a medical and paramedical anesthesia pair and supervised by simulation trainers.

Stress and resilience measures will be taken at various times during the study. Participants will be debriefed at the end of the simulation.

The primary objective is to analyze the correlation between anesthesia professionals' resilience and measured stress.Secondary objectives are to study the association between: SDNN-measured stress and VAS-reported stress, age and SDNN-measured stress, CD RISC 10 resilience and PSS10-reported stress, CD RISC resilience and VAS-reported stress, the effect of experience on SDNN-measured stress, multiple correlation of the different secondary criteria.

secondary criteria.

ELIGIBILITY:
Inclusion Criteria:

- volunteer in anesthesia

Exclusion Criteria:

* Rhythm disorders
* Endocrine pathology
* High blood pressure
* Pregnancy or breastfeeding in progress
* Taking anti-inflammatory or psychotropic drugs that interfere with the heart rate
* Interruption of professional practice in anesthesia > 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anaesthetic teams composed with :
  * 1 resident in anaesthesiology and critical care OR Anesthesiologist AND
  * 1 anaesthetic nursing student OR 1 anaesthetic nurse graduated
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-06-18 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | during the laryngospasm (during 3 minutes at 6 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Resilience | 5 days before scenario
  Measurement of resilience by Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40) in participants. A high score indicates better resilience.

SECONDARY OUTCOMES:
Self-reported stress | 5 days before scenario
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Self-reported stress | just Before the scenario (at 0 minute )
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Self-reported stress | just after briefing (at 3 minutes)
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Self-reported stress | just after the end of scenario (at 9 minutes)
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Self-reported stress | just after the debriefing (at 30 minutes)
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Perceived Stress Scale | 5 days before scenario
  The Perceived Stress Scale (PSS10 from 10 To 50) measures the degree to which respondents feel their lives are unpredictable, uncontrollable, and overloaded. A high score indicates more stress.
Age of anesthesia professionals | 5 days before scenario
  Age of anesthesia professionals: (quantitative variable)
Experience in anesthesia: | 5 days before scenario
  Experience in anesthesia: number of years since the beginning of specialized training training (quantitative variable)
Pediatric experience: | 5 days before scenario
  Pediatric experience: qualitative variable (yes, no)
Pediatric laryngospasm experience | 5 days before scenario
  Pediatric laryngospasm experience: qualitative variable: (yes, no)
Heart rate variability | 5 days before scenario (during 3 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Heart rate variability | Before the scenario (during 3 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Heart rate variability | during briefing (during 3 minutes at 0 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Heart rate variability | during the scenario before the laryngospasm (during 3 minutes at 3 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Heart rate variability | during the debriefing (3 minutes at 9 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants
Heart rate variability | after the debriefing (3 minutes at 30 minutes)
  Standard deviation of the average of RR intervals (SDNN in milliseconds) in participants

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Zafiriou, Principal Investigator — University Hospital, Grenoble; Julien Picard, M.D, Ph.D., Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France